CLINICAL TRIAL: NCT06935487
Title: Clinical Validation of Transrectal Multiparametric Ultrasound (PCaVision) for Detecting Clinically Significant Prostate Cancer: A European Head-to-Head Comparison With MRI in Primary Diagnosis and Active Surveillance Populations
Brief Title: European Multicenter Validation of PCaVision: A Head-to-Head Diagnostic Accuracy Study Comparing Multiparametric Transrectal Ultrasound to MRI for Clinically Significant Prostate Cancer Detection
Acronym: PCaVISTA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Angiogenesis Analytics (Industry)
Responsible Party: Principal Investigator, Harrie P. Beerlage, Prof. Dr. H.P. Beerlage, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL87353.000.24
Record Dates: First submitted 2025-04-04; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate biopsy; prostate biopsies; artificial intelligence; computer-aided diagnosis; magnetic resonance imaging; targeted biopsy; ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study uses a fully paired design, where each participant undergoes both interventions - PCaVision and MRI imaging - and receives biopsies based on each modality within the same study period.
Who Masked: Outcomes Assessor
Masking Description: Masking of Image Interpreters and Outcome Assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCaVision Imaging + PCaVision-Targeted Biopsy (Experimental): Participants undergo 3D multiparametric ultrasound (mpUS) imaging using PCaVision, a software-assisted diagnostic tool that combines B-mode, Shear Wave Elastography, and Contrast-Enhanced Ultrasound (CEUS).
  Suspicious lesions identified by PCaVision will be targeted for biopsy (up to 2 lesions, 3 cores each).
  * Transrectal 3D mpUS using PCaVision software (v1.1)
  * Injection of ultrasound contrast agent (SonoVue)
  * Targeted biopsy based on PCaVision lesion detection (up to 6 cores total)
  Interventions: Diagnostic Test: transrectal ultrasound of prostate (TRUS) with AI software algorithm
- MRI Imaging + MRI-Targeted Biopsy (Active Comparator): Participants undergo multiparametric MRI (mpMRI) of the prostate using 1.5T or 3T MRI systems.
  Suspicious lesions identified by MRI will be targeted for biopsy (up to 2 lesions, 3 cores each).
  * Prostate mpMRI with or without contrast
  * Image analysis following PI-RADS criteria
  * Targeted biopsy based on MRI lesion detection (up to 6 cores total)
  Interventions: Diagnostic Test: MRI prostate

INTERVENTIONS:
Diagnostic Test: transrectal ultrasound of prostate (TRUS) with AI software algorithm — Transrectal ultrasound of prostate (TRUS) with AI software algorithm for detection of lesions suspected for prostate cancer
  Arms: PCaVision Imaging + PCaVision-Targeted Biopsy
Diagnostic Test: MRI prostate — MRI for detection of lesions suspected for prostate cancer
  Arms: MRI Imaging + MRI-Targeted Biopsy

SUMMARY:
The goal of this clinical trial is to learn if a new ultrasound-based imaging method (PCaVision) can accurately detect clinically significant prostate cancer in adult men (18 years and older) who are either undergoing initial evaluation or are already in active surveillance for prostate cancer. The main questions it aims to answer are:

* Does PCaVision detect clinically significant prostate cancer as accurately as MRI?
* Can some men safely avoid prostate biopsies based on PCaVision imaging results?

Researchers will compare PCaVision-guided biopsies to MRI-guided biopsies to see if PCaVision performs as well as MRI in identifying aggressive prostate cancers.

Participants will:

* Undergo both an MRI and a PCaVision ultrasound scan
* Receive targeted prostate biopsies based on any suspicious areas found in either scan
* Possibly have follow-up visits to monitor for biopsy-related side effects

DETAILED DESCRIPTION:
Rationale The incidence of prostate cancer (PCa) has increased over the years. To diagnose PCa, histopathological confirmation is required. Different diagnostic pathways are currently available. Systematic biopsies have long been the cornerstone in the diagnostic work-up of men suspected of prostate cancer. However, systematic biopsies can lead to under-diagnosis of clinically significant prostate cancer (csPCa), and each biopsy is associated with the risk of infection and other side effects.

In the magnetic resonance imaging (MRI) pathway, targeted biopsies are only performed when suspicious lesions are detected on MRI. The MRI pathway purposely detects fewer clinically insignificant prostate cancers (ciPCa), but has an increased sensitivity for csPCa and improved localization accuracy of suspicious regions. The MRI-based strategy is now recommended as the first-line investigation. However, reported sensitivities and specificities for MRI vary widely between studies, which can be attributed to differences in MRI equipment, study design, reference standard quality, and inter-observer variability. Moreover, MRI has limited availability and is a time-consuming and expensive imaging modality.

Transrectal ultrasound (TRUS), which is widely available, more cost-effective, and familiar to urologists, may offer a valid alternative. In an ultrasound-based diagnostic pathway, 3D contrast-enhanced ultrasound (CEUS) combined with contrast ultrasound dispersion imaging (CUDI) focuses on detecting angiogenetic changes in the microvascular architecture to localize lesions suspicious for PCa, followed by targeted biopsies for histological confirmation.

PCaVision is a software package designed to support the diagnosis of csPCa by integrating 3D B-mode, 3D Shear Wave Elastography (SWE), and 4D CEUS scans. The PCaVision algorithm was trained on a cohort of 252 patients using prostatectomy pathology as the reference standard, and 83 "negative" patients (no suspicious MRI lesions or positive prostate biopsies). Internal validation showed a sensitivity and specificity of 0.82 and 0.82, respectively. These results led to a first prospective clinical investigation in the Netherlands to demonstrate non-inferiority compared to the MRI-based pathway (NCT06281769). That initial prospective trial aimed to compare the two diagnostic pathways in biopsy-naïve patients under tightly controlled conditions (e.g., 3T MRI, transperineal biopsies, and cognitive or fusion targeting using MIM software). These conditions, however, are not generalizable across Europe, where 1.5T and 3T MRI are used interchangeably, both transperineal and transrectal biopsy approaches are employed, and various fusion systems are in use. Additionally, the previous study excluded patients in active surveillance (AS) and those with prior negative biopsies, who represent a substantial portion of the demand for PCa diagnosis and biopsy guidance.

The objective of the European head-to-head trial described in this protocol is to compare the diagnostic accuracy of two different imaging pathways for detecting csPCa in a broader, more generalizable European setting: (1) the PCaVision-targeted biopsy pathway and (2) the MRI-targeted biopsy pathway. The trial aims to demonstrate the non-inferiority of the PCaVision pathway compared to the MRI pathway in two cohorts: (1) biopsy-naïve and prior negative patients and (2) patients undergoing active surveillance. A fully paired design will be used. The updated PCaVision version 1.1 will be employed in this study, incorporating enhancements to reduce unusable scans and improve diagnostic accuracy and user experience.

Objective

The primary objective is to demonstrate the non-inferiority of csPCa detection in targeted biopsies guided by PCaVision imaging (PCaVision pathway) compared to targeted biopsies guided by MRI (MRI pathway) in two distinct patient cohorts:

1. Biopsy-naïve and prior-negative patients
2. Patients under active surveillance (AS) Clinically significant PCa (csPCa) is defined as International Society of Urological Pathology (ISUP) Grade Group (GG) ≥ 2 in any biopsy core obtained from a lesion.

The secondary objectives include:

1. Comparing the proportion of participants in whom targeted biopsies could be safely omitted in the PCaVision pathway versus the MRI pathway. Safe omission is defined as no lesions identified for targeted biopsy by PCaVision and no csPCa detected by MRI-targeted or systematic biopsies.
2. Conducting the same diagnostic comparison across different definitions of csPCa, including:

   * ISUP ≥ 3
   * ISUP ≥ 2 with cribriform growth and/or intraductal carcinoma (CR/IDC)
   * ISUP = 1
3. Comparing the number of participants for whom PCaVision or MRI produced insufficient image quality.
4. Calculating csPCa detection rates across specific subgroups:

   * Men treated with 5-alpha reductase inhibitors (5-ARI) for ≥3 months
   * Men with a history of prostate surgery for lower urinary tract symptoms (LUTS)
   * Biopsy-naïve and prior-negative patients excluding those under 5-ARI treatment or with prostate surgery history
   * AS patients excluding those under 5-ARI treatment or with prostate surgery history Study Design This is a prospective, diagnostic accuracy study using a fully paired design. Study Population The study will include men aged 18 years or older who are scheduled for prostate MRI due to either a suspicious digital rectal examination (DRE) and/or elevated PSA, or as part of routine active surveillance follow-up.

Intervention

All participants will undergo both:

* 3D multiparametric ultrasound (mpUS) imaging using PCaVision
* Multiparametric MRI Suspicious lesions will be identified independently on each modality. If lesions are detected, targeted biopsies will be performed based on the findings.

Biopsy procedure:

* If one lesion is detected: 3 targeted biopsies
* If two lesions: 3 biopsies per lesion (6 total)
* If three or more lesions: 2 selected lesions will be biopsied (3 biopsies per lesion)

Selection criteria:

* For MRI: PI-RADS score and lesion size
* For PCaVision: predicted csPCa probability and lesion size A maximum of 6 biopsies per imaging technique will be performed (maximum 12 study-driven biopsies per participant). This does not include systematic biopsies, which may be conducted according to the standard of care at the participating center. All biopsies will be conducted during a single visit.

Main Study Endpoint The primary endpoint is the detection of clinically significant prostate cancer (GG ≥ 2) based on histopathological examination of targeted biopsies. The study aims to demonstrate that detection using the PCaVision pathway is not inferior to detection using the MRI pathway within a predefined non-inferiority margin of 5 percentage points for both patient cohorts.

Burden, Risks, and Benefits In most participating centers, current clinical care involves MRI-targeted and possibly systematic biopsies. These care practices will remain unchanged in the study. Systematic biopsies are not part of the formal head-to-head comparison between MRI and PCaVision.

Potential benefits to participants include detection of additional cancers that MRI may miss. Broader study results may help expand access to effective diagnostic imaging, especially in settings with limited MRI availability.

Additional targeted biopsies may be required based on PCaVision findings, which carry minor risks such as infection or bleeding. The use of ultrasound contrast agent may pose minimal and rare risks, typically transient and mild. Overall, the burden and risk associated with participation are considered low.

ELIGIBILITY:
Inclusion criteria:

1. male
2. 18 years of age or older
3. scheduled for evaluation by prostate MRI due to:

   * suspicious digital rectal examination (DRE) and/or
   * Elevated serum PSA levels, or as part of active surveillance (AS) follow-up
4. Have provided written informed consent

Exclusion criteria:

1. Active urinary tract infection or prostatitis
2. A history of cardiac right-to-left shunt
3. Allergy to sulphur hexafluoride or any other ingredient in the ultrasound contrast agent SonoVue
4. Current treatment with dobutamine
5. Severe pulmonary hypertension (pulmonary artery pressure > 90 mmHg), uncontrolled systemic hypertension, or respiratory distress syndrome
6. Any other contraindication to MRI or 3D mpUS imaging
7. Inability to understand the language of the patient information (i.e., language barrier)
8. Previous treatment with focal therapy for prostate cancer (e.g., HIFU, cryotherapy, laser ablation, etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Clinically Significant Prostate Cancer (csPCa) Detected by PCaVision-Targeted Biopsies Compared to MRI-Targeted Biopsies | 12 months
  Clinically significant prostate cancer (csPCa) is defined as ISUP Grade Group (GG) ≥ 2. The number of participants in whom csPCa is detected through PCaVision-targeted biopsies will be compared to the number of participants with csPCa detected through MRI-targeted biopsies. The comparison will be performed separately for two patient cohorts:
  1. Biopsy-naïve or prior negative biopsy patients
  2. Patients under active surveillance (AS) A non-inferiority margin of 5 percentage points will be used.

SECONDARY OUTCOMES:
Number of Participants With No Suspicious Lesions on PCaVision and No Clinically Significant Prostate Cancer (csPCa) Detected by MRI-Targeted or Systematic Biopsies | 12 months
  This outcome measures the number of participants for whom PCaVision did not identify any suspicious lesions and in whom no csPCa (ISUP Grade Group ≥ 2) was subsequently found on MRI-targeted or systematic biopsies. The purpose is to evaluate the potential for safely omitting biopsies when PCaVision imaging does not indicate suspicion of csPCa. Data will be reported as a count and proportion of participants meeting this criterion.
Number of Participants With Prostate Cancer Detected by PCaVision or MRI According to Alternative Definitions of Clinically Significant Cancer | 12 months
  This outcome measures the number of participants in whom prostate cancer is detected through PCaVision-targeted or MRI-targeted biopsies using three different histopathological definitions:
  * ISUP Grade Group ≥ 3
  * ISUP Grade Group ≥ 2 with cribriform growth and/or intraductal carcinoma (CR/IDC)
  * ISUP Grade Group = 1
  The data will be reported as the number and proportion of participants in each category for both imaging pathways.
Number of Participants With Insufficient Image Quality for Diagnostic Assessment on PCaVision or MRI | 12 months
  This outcome measures the number of participants for whom the image quality of either PCaVision or MRI was rated as insufficient to allow for a diagnostic assessment. Insufficient quality is defined per site-specific criteria or based on the inability to identify or evaluate prostate lesions using the imaging modality. Data will be reported as the number and proportion of participants with insufficient image quality for each imaging technique.
Number of Participants With Clinically Significant Prostate Cancer (csPCa) Detected in Prespecified Subgroups | 12 months
  This outcome measures the number and proportion of participants with csPCa (ISUP Grade Group ≥ 2) detected through targeted biopsies (PCaVision and/or MRI) within the following subgroups:
  * Participants treated with 5-alpha reductase inhibitors (5-ARI) for ≥ 3 months
  * Participants with a history of prostate surgery for lower urinary tract symptoms (LUTS)
  * Biopsy-naïve or prior-negative participants excluding those treated with 5-ARI or with prior surgery
  * Active surveillance (AS) participants excluding those treated with 5-ARI or with prior surgery
  Detection rates will be compared across these subgroups for each imaging pathway.

CONTACTS AND LOCATIONS:
Overall Officials: dr. Oddens, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (10):
- France (2):
  - Institut Paoli- Calmettes, Marseille
  - L'Institut Mutualiste Montsouris, Paris
- Germany (3):
  - University Klinikum Bonn, Bonn
  - Martini-Klinik am UKE, Hamburg
  - Urologische Klinik München- Planegg, Planegg
- Italy (2):
  - Università degli Studi di Foggia, Foggia
  - University of Padua, Padua
- Amsterdam UMC, Amsterdam, Netherlands
- Oslo University hospital Ullevål, Oslo, Norway
- Fundació Puigvert, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing Statement Section
  * Plan to Share IPD: Yes
  * Plan Description:
  De-identified individual participant data (IPD) will be shared with qualified researchers after the main study results are published. Data sharing will be governed by a data use agreement and ethical approvals.
  • IPD Description:
  The following individual-level data will be shared:
  * Participant demographics (e.g., age, PSA level, clinical cohort)
  * Imaging results from PCaVision and MRI (e.g., lesion scores, heatmaps, image quality)
  * Histopathological biopsy outcomes (e.g., ISUP Grade Group, csPCa status)
  * Subgroup classifications (e.g., use of 5-ARI, prior prostate surgery)
  * Imaging quality and adverse events (de-identified)
    • Supporting Documents:
  * Study Protocol
  * Statistical Analysis Plan (SAP)
  * Informed Consent Form (ICF) [if permitted] • Time Frame: Data will become available after publication of the primary results and completion of the trial, estimated to be around March 2026. Data will remain avail
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after publication of the primary results and completion of the trial, estimated to be around March 2026. Data will remain available for at least 5 years thereafter.
Access Criteria: Data will be shared with qualified researchers affiliated with academic institutions or non-profit organizations. Requests must include a methodologically sound proposal and will require a data use agreement.

REFERENCES:
- [Background] Jager A, Vilanova JC, Michi M, Wijkstra H, Oddens JR. The challenge of prostate biopsy guidance in the era of mpMRI detected lesion: ultrasound-guided versus in-bore biopsy. Br J Radiol. 2022 Mar 1;95(1131):20210363. doi: 10.1259/bjr.20210363. Epub 2021 Jul 29. PMID 34324383
- [Background] van Moorselaar RJ, Voest EE. Angiogenesis in prostate cancer: its role in disease progression and possible therapeutic approaches. Mol Cell Endocrinol. 2002 Nov 29;197(1-2):239-50. doi: 10.1016/s0303-7207(02)00262-9. PMID 12431818
- [Background] van den Kroonenberg DL, Jager A, Garrido-Utrilla A, Reitsma JB, Postema AW, Beerlage HP, Oddens JR. Clinical Validation of Multiparametric Ultrasound for Detecting Clinically Significant Prostate Cancer Using Computer-Aided Diagnosis: A Direct Comparison with the Magnetic Resonance Imaging Pathway. Eur Urol Open Sci. 2024 Jul 1;66:60-66. doi: 10.1016/j.euros.2024.06.012. eCollection 2024 Aug. PMID 39050912
- [Background] Jager A, Zwart MJ, Postema AW, van den Kroonenberg DL, Zwart W, Beerlage HP, Oddens JR, Mischi M. Development and validation of a framework for registration of whole-mount radical prostatectomy histopathology with three-dimensional transrectal ultrasound. BMC Urol. 2025 Apr 3;25(1):73. doi: 10.1186/s12894-025-01736-4. PMID 40175990